CLINICAL TRIAL: NCT02278848
Title: Multimodal Investigation in the Diagnosis and Treatment of Chronic Adult Hydrocephalus
Acronym: Multimod'HCA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PHAO 2013- KM / Multimod'HCA
Record Dates: First submitted 2014-07-18; First posted 2014-10-30 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2023-01

CONDITIONS: Chronic Adult Hydrocephalus
Keywords: Computerised gait analysis; Ultrasound measurement of cerebral pulsatility; MRI flow; Urinary incontinence scale; Subtractive lumbar puncture
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Diagnosis of ICAH (Experimental): One arm: patients with chronic adult hydrocephalus.
  All patients have: Computerised gait analysis, Ultrasound measurement of cerebral pulsatility, MRI flow, Urinary incontinence scale
  Interventions: Other: Diagnosis of ICAH using new investigative techniques (computerised gait analysis, ultrasound, MRI flow, urinary incontinence scale)

INTERVENTIONS:
Other: Diagnosis of ICAH using new investigative techniques (computerised gait analysis, ultrasound, MRI flow, urinary incontinence scale) — Diagnosis of ICAH using new investigative techniques (computerised gait analysis, ultrasound, MRI flow, urinary incontinence scale)

SUMMARY:
Idiopathic chronic adult hydrocephalus (ICAH) is due to expansion of the fluid-filled cavities in the brain. The clinical symptoms are gait disturbance, mental decline and incontinence. Treatment involves installing a ventriculoperitoneal shunt which is known to be able to induce regression of the symptoms in many cases meaning that ICAH is a classic, curable cause of dementia. Diagnosis relies on comparing symptoms before and after depleting cerebrospinal fluid (CSF) via a lumbar puncture (LP). In practice, the situation is complicated: improvement is often incomplete and there is no consensus on either how to assess the symptoms or how they change after CSF depletion. In consequence, the decision whether not to undertake surgery often depends on the neurosurgeon's clinical impression.

Over recent years, the cognitive profile of patients with ICAH has become better characterised and reproducible, objective techniques have been developed to assess motor function and CSF flow in the brain.

The investigators project aims to define the value of these new investigative techniques in the positive diagnosis of ICAH, in comparison to current decision-making tools.

ELIGIBILITY:
Inclusion Criteria:

* Adult 65 years or older
* Hospitalized patients (at the University Hospital of Tours) requiring the assessment of chronic hydrocephalus in adults, suspected clinically
* Patient undergoing Lumbar Puncture subtractive
* Informed consent form signed
* Affiliated to a medical insurance

Exclusion Criteria:

* Contraindications to MRI
* Inability to walk or to stand before having lumbar puncture
* Patient under trusteeship and guardianship, or judicial protection

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-07-21 (Actual); Primary Completion 2018-07-21 (Actual); Study Completion 2018-07-21 (Actual)

PRIMARY OUTCOMES:
Cerebrospinal fluid biomarkers of degeneration from Alzheimer's disease. | 5 days
  Association between the decision-making with regard to permanent CSF shunt and the response to subtractive lumbar puncture
Computerised gait analysis | 5 days
  Association between the decision-making with regard to permanent CSF shunt and the Computerised gait analysis,
Ultrasound measurement of cerebral pulsatility | 5 days
  Association between the decision-making with regard to permanent CSF shunt and the Ultrasound measurement of cerebral pulsatility,
Qualitative and quantitative analysis (average speed and flow) of the hydrodynamic characteristics of the cerebrospinal fluid. | 5 days
  Association between the decision-making with regard to permanent CSF shunt and the MRI flow,
Urinary incontinence | 5 days
  Association between the decision-making with regard to permanent CSF shunt and the Urinary incontinence scale

CONTACTS AND LOCATIONS:
Overall Officials: Karl MONDON, Principal Investigator — CHRU de Tours
Locations (1):
- CHRU de Tours, Tours, France